CLINICAL TRIAL: NCT03961737
Title: Study of the Response to Irradiation on Prostatic Explants ex Vivo, as a Predictive Factor of the Clinical Response to Irradiation of Prostate Cancers
Acronym: EXPLANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-N-2016-05
Record Dates: First submitted 2019-05-15; First posted 2019-05-23 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
Keywords: radiotherapy; explants; transcriptomic; immunohistochemistry
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prostatic explants (Experimental): A first series of biopsies will be performed during the procedure to place the gold grains prior to radiotherapy. Explants will be performed from these biopsies. Half of these explants will be irradiated with a research irradiator at a dose of 2 Gy then placed for 24 hours in an appropriate culture medium. The other half will be directly cultured for 24 hours. After 24 hours of incubation, half of the irradiated explants and half of the explants will be used to study the transcriptome. The tissues will be stored in RNAlater solution and then frozen at -80°C. The remaining half explants will be used for immunohistochemical analysis. Two years after the end of radiotherapy, a new series of biopsies will be performed for research, in order to verify histologically the effectiveness of radiotherapy.
  Interventions: Procedure: prostate biopsies

INTERVENTIONS:
Procedure: prostate biopsies — Before radiotherapy treatment, prostate biopsies will be performed in each patient. From these biopsies, explants will be performed. Half of these explants will be irradiated ex vivo and the other half will not receive any prior treatment.
  Then the patient will receive radiotherapy. It will be reviewed 2 years after the end of radiotherapy. New prostate biopsies will be performed to evaluate the tumor response to radiotherapy and to characterize the immunohistochemical and transcriptomic profiles of non-responder patients.

SUMMARY:
Of the 50,000 prostate cancers that occur each year in France, more than half will benefit from curative radiotherapy, alone or in combination with hormone therapy from 6 months to 3 years depending on the stage of the disease. At present, there are few ways to predict the response to this irradiation.

Evaluating the early response of tumor tissue to irradiation could predict the final response to treatment. It is difficult to offer biopsies during treatment for reasons of patient comfort. This is why this study consists in analysing transcriptomic and protein responses (immunohistochemistry) to irradiation on ex vivo prostate explants. These explants will be irradiated after culture and the transcriptional and immunohistochemical changes analysed before and after irradiation to determine an early tumor tissue response profile to irradiation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Patient with non-operated prostate adenocarcinoma for whom radiotherapy treatment is scheduled
3. Signed Informed Consent
4. No contraindications to biopsy performance:

   * No anticoagulant treatment in progress
   * Absence of infection during diagnostic biopsies
   * Absence of pain requiring level 2 analgesics during diagnostic biopsies
   * Absence of bleeding complications during diagnostic biopsies
   * Absence of anal stenosis
5. Normal coagulation examination :

   * Prothrombin Ratio between 80 and 100%.
   * Active Cephalin Time from 24 to 41 seconds, > 1.5 times that of the indicator
   * Platelets > 150,000 G/L
   * International Normalised Ratio(INR) = 1 after stopping the anticoagulant
6. No contraindication to MRI:

   * Ocular metallic foreign body
   * Pacemaker
   * Old mechanical heart valve
   * Ancient vascular clips on cranial aneurysms

Exclusion Criteria:

1. History of radical prostatectomy. A history of transurethral prostate resection is not a contraindication
2. History of prostate infection
3. Hemorrhagic complications in diagnostic biopsies
4. Pain requiring level 2 analgesics in diagnostic biopsies
5. Anticoagulant treatment in progress (aspirin will be stopped 1 week before biopsies are performed)
6. Abnormal coagulation assessment
7. Anal stenosis
8. Contraindications to radiotherapy: chronic inflammatory bowel disease, scleroderma
9. Protected or tutored patient
10. Patient whose follow-up at two years is not possible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
biopsy tumor response | 24 months after radiotherapy
  The centralized anatomopathological study of prostate biopsies will classify patients into good responders (absence of viable tumour cells) and poor responders (persistence of viable tumour cells).

SECONDARY OUTCOMES:
Change in Biochemical response to radiotherapy. | every 6 months for a maximum total of 24 months
  Biological response to radiotherapy the biological response to radiotherapy is assessed by measuring serum PSA levels according to Phoenix criteria, nadir 2 ng/ml
prostatic Magnetic Resonance Imaging | 24 months after radiotherapy
  Prostate MRI 2 years after the end of radiotherapy, used to identify the area affected by the tumor

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane SUPIOT, MD, Principal Investigator — ICO
Locations (1):
- ICO, Saint-Herblain, France